CLINICAL TRIAL: NCT01715506
Title: Modeling and Evaluating Evidence Based Continuing Education in Nursing Home Dementia Care
Brief Title: Continuing Education in Nursing Home Dementia Care
Acronym: MEDCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bergen University College (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Frode F. Jacobsen, Professor, Director, Bergen University College
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2012/304
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Dementia; Agitation
Keywords: Dementia; Resident; Nursinghome; Use of restraint; Agitation
MeSH Terms: conditions — Dementia; Psychomotor Agitation | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Educational intervention (Experimental): Educational intervention with two days of lecture/course for the whole staff in the selected department in each nursing home and six monthly sessions of counselling in smaller groups
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Educational intervention — The educational intervention (EI), Relation Related Care (RRC), consists of a two-day seminar and one hour monthly guidance for six months. Course material, a book particularly designed for this intervention and dealing with person centered care and use of restraint, is distributed ahead of the course part of the intervention to all participants.

SUMMARY:
This is a single-blinded controlled cluster-randomized intervention trial recruiting staff from 24 NHs in three counties in the region of Western Norway, randomly selected from the total NH population in the region. A cluster is defined as a working ward of a larger NH, without shared facilities or staff. The 24 NHs are randomized into two groups, for intervention (12) and control (12). One department in each is selected for intervention and data collection will take place also in one department in each of the NHs in the control group. Hence the analyzed units (clusters) are NH departments. The educational intervention (EI), Relation Related Care (RRC), consists of a two-day seminar and one hour monthly guidance for six months. A seven-month educational intervention will be performed, and due to ethical issues the control group will receive the same intervention after the second follow-up. Effects will be measured on resident and care staff level at baseline before randomization, after the intervention (7 months) and at follow-up (7 months later) of the intervention group.

DETAILED DESCRIPTION:
Purpose:

Dementia is a major challenge for our society. In Norway, around 40 % of persons suffering from dementia live in nursing homes (NH), and the majority experiences severe functional impairments and complex needs including associated behavioral changes. International studies indicate that NH residents with cognitive impairment and high dependency are most likely to be restrained physically. There is evidence of various adverse effects such as injuries, reduced psychological well-being or decreased mobility related to the use of physical restraint. Moreover, in addition to ethical and professional arguments, there is evidence supporting that user-involvement and shared decision-making have positive effects for both residents and staff. The aim of the present study (MEDCED) is to carry out an educational intervention in care staff to test its potential effect on use of restraint in NH residents with dementia and increase job-satisfaction in care staff.

Description:

This is a single-blinded controlled cluster-randomized intervention trial recruiting staff from 24 NHs in three counties in the region of Western Norway, randomly selected from the total NH population in the region. A cluster is defined as a working ward of a larger NH, without shared facilities or staff. The 24 NHs are randomized into two groups, for intervention (12) and control (12). One department in each is selected for intervention and data collection will take place also in one department in each of the NHs in the control group. Hence the analyzed units (clusters) are NH departments. The educational intervention (EI), Relation Related Care (RRC), consists of a two-day seminar and one hour monthly guidance for six months. A seven-month educational intervention will be performed, and due to ethical issues the control group will receive the same intervention after the second follow-up. Effects will be measured on resident and care staff level at baseline before randomization, after the intervention (7 months) and at follow-up (7 months later) of the intervention group.

An analysis of how many units needs to be included are based on 12+12 clusters. Two calculations have been performed. The first calculation is based on how big is the reduction in use of restraints. We assume in our model that there will be a 60 % reduction in use of restraints in the intervention group and 33 % reduction in the control group (Hawthorne effect). For this reason we need to include averagely 13 patients in each department/unit in order to achieve a statistical power of 0,8.

Measures on resident will be collected by a skilled research nurse blind to the study. Care staff measures will be collected through a questionnaire distributed directly to the care staff, provided with a stamped envelope to return the questionnaire directly to the research group. In addition, department characteristics (like type of department, staff coverage, architecture) will be registered.

A research team will lead the EI, and four facilitator teams each consisting of one nurse and one assistant professor from a nursing schools will be responsible for the EI of the decision-making model in the NHs. The Educational intervention will be carried out in two steps, firstly from researchers to the educators (EI 1) and secondly from the educators to the NH staff (EI 2)

ELIGIBILITY:
Inclusion Criteria:

* Dementia

Exclusion Criteria:

* non-dementia

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Restraint change | Assessment in 6-8 months, publication in approximately 18-20 months
  Use of restraint be assessed by a trained research assistant, employing a form specifically developed for this project, assessing use of restraint.

SECONDARY OUTCOMES:
Psychotropic drug change | Assessment in 6-8 months, publication in approximately 18-20 months
  Use of psychotropic drugs will be assessed by a trained research assistant, registering the total medication of the patients from the patient chart.

CONTACTS AND LOCATIONS:
Overall Officials: Frode F Jacobsen, PhD, Study Director — Bergen University College
Locations (24):
- Norway (24):
  - Flora Omsorgssenter, Florø, Flora
  - Furuhaugane Omsorgssenter, Florø, Flora
  - Solas bo- og rehabiliteringssenter, Ålgård, Gjesdal
  - Husnestunet, Rosendal, Kvinnherad
  - Rosendalstunet, Rosendal, Kvinnherad
  - Kvitsoy kombisenter, Stavanger, Kvitsoy
  - Luster Sjukeheimsteneste, avd. Gaupne, Sogndal, Luster
  - Samnangerheimen, Bergen, Samnanger
  - Ask bo- og omsorgssenter, Askoy
  - Stiftelsen Nykirkehjemmet, Bergen
  - Landaas Meninghets Eldresenter, Bergen
  - Midtbygda sykehjem, Bergen
  - Teiglandshagen bufellesskap, Bømlo
  - Bygdaheimen, Eidfjord
  - Gulen Sjukeheim, Gulen
  - Laerdal Alders- og Sjukeheim, Lærdal
  - Roldal pleie og omsorgstjeneste, Odda
  - Byhagen Bo og Aktivitetssenter, Sandnes
  - Sogndal Omsorgssenter, Sogndal
  - Bergåstjern Sykehjem, Stavanger
  - Boganes Bokollektiv, Stavanger
  - Oyane Sykehjem, Stavanger
  - Tysnes Sjukeheim, Tysnes
  - Tysvaertunet, Tysvær

REFERENCES:
- [Derived] Jacobsen FF, Mekki TE, Forland O, Folkestad B, Kirkevold O, Skar R, Tveit EM, Oye C. A mixed method study of an education intervention to reduce use of restraint and implement person-centered dementia care in nursing homes. BMC Nurs. 2017 Sep 18;16:55. doi: 10.1186/s12912-017-0244-0. eCollection 2017. PMID 28936121